CLINICAL TRIAL: NCT02202369
Title: Multimodal Analgesia vs. Routine Care Pain Management for Lumbar Spine Fusion Surgery: A Prospective Randomized Study
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment and subject followup rates
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Charlotte Orthopedic Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9080
Record Dates: First submitted 2014-07-14; First posted 2014-07-29 (Estimated); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Single Level Lumbar Decompression and Fusion Spine Surgery
Keywords: Multimodal Analgesia; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodal Analgesia (MMA) Treatment (Experimental)
  Interventions: Other: Multimodal Analgesia Treatment
- Standard of Care Pain Managment Protocol (Active Comparator)
  Interventions: Other: Standard of Care Pain Management Protocol

INTERVENTIONS:
Other: Multimodal Analgesia Treatment — Subjects are given medications preop (Pregabalin, Oxycodone, Acetaminophen, Transdermal Scopolamine, Cyclobenzaprine), intraop (Propofol induction, Sevoflorane maintenance, Dexamethasone, Fentanyl, Ketamine, Marcaine, Zofran) and postop(Acetaminophen, Pregabalin, Tramadol, Cyclobenzaprine) that implement a multi-modal approach to managing pain.
  Arms: Multimodal Analgesia (MMA) Treatment
Other: Standard of Care Pain Management Protocol — Subjects will be treated with patient controlled (standard of care) narcotic analgesia for pain management. (Marcaine, Dexamethasone, Zofran, Morphine, Acetaminophen, Cyclobenzaprine)
  Arms: Standard of Care Pain Managment Protocol

SUMMARY:
The purpose of this study is to determine if post-operative pain and rate of recovery are improved in patients undergoing spine surgery using MMA (multimodal analgesia) compared to usual analgsic care.

DETAILED DESCRIPTION:
Specific Aim #1: To compare the postoperative pain levels of single level lumbar fusion patients treated with either MMA pain management protocol or standard pain management protocol.

Controlling postoperative pain is a critical first step in facilitating a patient's recovery and improved quality of life. In-hospital pain levels will be measured using a numeric pain scale on a scale of 0-10. Pain assessment is conducted by the hospital nurses as a standard of care protocol. Assessments are every four to six hours, within 60 minutes after receiving a pain medication

Hypothesis: Patients treated with the MMA pain protocol will have significantly less immediate postoperative pain as compared to patients treated with the standard pain protocol.

Specific Aim #2: To compare the immediate postoperative, or in-hospital, narcotic consumption of single level lumbar fusion patients treated with either MMA pain management protocol or standard pain management protocol.

Decreasing narcotic consumption following lumbar spinal fusion surgery is important for faster recovery for the patient, decreasing narcotic related side effects (nausea and vomiting, lethargy, ileus, etc) as well as lowering overall treatment costs. The total amount of narcotic use during the course of the hospitalization for each subject will be recorded. Dosages of narcotics will be converted to morphine equivalents.

Hypothesis: Patients treated with the MMA pain protocol will consume significantly less immediate postoperative narcotic pain medications compared to patients treated with the standard pain protocol.

Specific Aim #3: To compare the length of hospital stay of single level lumbar fusion patients treated with either MMA pain management protocol or standard pain management protocol.

Decreasing the amount of time patients remain in the hospital may decrease the time it takes a patient to return to personal and societal responsibilities. Additionally it reduces the patients risk of a nosocomial infection and reduces the costs of the surgery.

Hypothesis: Patients treated with the MMA pain protocol will have a significantly reduced length of stay in the hospital compared to patients treated with the standard pain protocol.

Specific Aim #4: To compare postoperative quality of life of single level lumbar fusion patients treated with either MMA pain management protocol or standard pain management protocol.

The primary purpose of lumbar fusion surgery is to improve the quality of life for patients. The Oswestry Disability Index (ODI) will be used as a disease specific measure. The Veterans Rand 12 (VR-12) will be used as a general health outcome measure. Each of these patient reported outcome measures will be collected pre-operatively and at each of the following postoperative visits: 2 weeks, 6 weeks, 3 month, 6 visit, 1 visit, and 2 year.

Hypothesis: Patients treated with the MMA pain protocol will have significantly greater improvement in Quality of Life measures compared to patients treated with the standard pain protocol and this will be sustained out to two years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing a single level lumbar decompression and fusion
2. > 18 years of age and < 70 years of age
3. The subject is willing and able to understand, sign and date the study specific patient informed consent and HIPAA authorization to volunteer participation in the study

Exclusion Criteria:

1. Patients with liver disease (documented liver function test abnormality)
2. Patients with renal disease (documented glomerular filtration rate < 60mL/min/1.73m2)
3. Patients with a baseline (pre-operative) opioid use greater than 30 mg of morphine equivalents/day.
4. Patients with active alcohol dependence
5. Patients with active illicit drug dependence
6. Patients < 18 years of age and >70 years of age
7. Patients allergic to any medication given in either arm (list medications)
8. Patients who have a seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain level using a verbal numeric pain scale (NPS) | In hospital (participants will be followed for the duration of the hospital stay, an expected average of 2 days)
  While in the hospital, patient's pain is assessed by a nurse-driven standard of care protocol. Assessments are typically every four to six hours or within 60 minutes after receiving an intravenous or oral analgesic medication. This assessment includes rating subjective rating of ones pain on a verbal numeric rating scale (NRS) of 0-10. The maximum pain score for each post-operative day will be compared.

SECONDARY OUTCOMES:
Patient satisfaction | In hospital (participants will be followed for the duration of the hospital stay, an expected average of 2 days)
  As part of the nurse driven standard of care protocol, patients are asked if their pain level is acceptable during their stay in the hospital
Narcotic consumption | In hospital (participants will be followed for the duration of the hospital stay, an expected average of 2 days)
  The total amount of narcotic use during the course of hospitalization for each subject will be recorded. Dosages of narcotics will be converted to morphine equivalents
Length of stay | Hospital discharge (an expected average of 2 days after surgery)
  The number of hours of hospitalization from entering the recovery room (time zero) until the patient meets discharge criteria
Discharge destination | Hospital discharge (an expected average of 2 days after surgery)
  As standard of care this data point will be documented in the patients chart. It is categorized as patient home, rehabilitation facility, or skilled nursing facility
Oswestry Disability Index (ODI) | pre-operative, 2 week post-operative, 6 week post-operative, 3 month post-operative, 6 month post-operative, 1 year post-operative, 2 year post-operative
  A disease specific questionnaire
The Veterans Rand 12 (VR-12) | pre-operative, 2 week post-operative, 6 week post-operative, 3 month post-operative, 6 month post-operative, 1 year post-operative, 2 year post-operative
  A general health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alden Milam, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States